CLINICAL TRIAL: NCT03989466
Title: Phase Ib Pilot Study of Itacitinib With Alemtuzumab in Patients With T-Cell Prolymphocytic Leukemia (T-PLL)
Brief Title: Itacitinib and Alemtuzumab in Treating Patients With T-Cell Prolymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0054; NCI-2019-03203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0054 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Recurrent T-Cell Prolymphocytic Leukemia; T-Cell Prolymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic, T-Cell | interventions — Alemtuzumab; itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (itacitinib, alemtuzumab) (Experimental): CYCLE 1: Patients receive itacitinib PO QD on days 1-28 and alemtuzumab IV over 2 hours on days 15, 17, 19, 21, 23, 25, and 27 in the absence of disease progression of unacceptable toxicity.
  CYCLE 2 AND BEYOND: Patients receive itacitinib PO QD on day 1-28 and alemtuzumab IV over 2 hours on days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, and 27. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients who achieve a response (CR/CRi or PR) may receive itacitinib for up to 8 additional cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Alemtuzumab; Drug: Itacitinib

INTERVENTIONS:
Biological: Alemtuzumab — Given IV
  Other Names: Anti-CD52 Monoclonal Antibody; Campath; Campath-1H; LDP-03; Lemtrada; MabCampath; Monoclonal Antibody Campath-1H
Drug: Itacitinib — Given PO
  Other Names: INCB 039110; INCB-039110; INCB039110

SUMMARY:
This phase Ib trial studies the side effects and best dose of alemtuzumab when given together with itacitinib in treating patients with T-cell prolymphocytic leukemia. Itacitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with alemtuzumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving itacitinib and alemtuzumab may work better in treating patients with T-cell prolymphocytic leukemia compared to standard of care treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of itacitinib in combination with alemtuzumab in patients with T-cell prolymphocytic leukemia (T-PLL).

SECONDARY OBJECTIVES:

I. To evaluate the event free survival (EFS) in patients (pts) with T-PLL treated with itacitinib in combination with alemtuzumab.

II. To evaluate response complete remission (CR), complete remission without blood count recovery (CRi), or partial remission (PR) (CR/CRi or PR) of itacitinib in combination with alemtuzumab in patients with T-PLL.

III. To explore the single-agent activity of itacitinib in pts with T-PLL. IV. To assess the time to response, response duration, and overall survival (OS) in pts with T-PLL treated with the combination of itacitinib and alemtuzumab.

EXPLORATORY OBJECTIVES:

I. To explore the effect of itacitinib on STAT5 phosphorylation in pts with T-PLL II. To explore the association of pretreatment somatic mutations and the dynamics of STAT5 phosphorylation with response.

OUTLINE: This is a dose-escalation study of alemtuzumab.

CYCLE 1: Patients receive itacitinib orally (PO) once daily (QD) on days 1-28 and alemtuzumab intravenously (IV) over 2 hours on days 15, 17, 19, 21, 23, 25, and 27 in the absence of disease progression of unacceptable toxicity.

CYCLE 2 AND BEYOND: Patients receive itacitinib PO QD on day 1-28 and alemtuzumab IV over 2 hours on days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, and 27. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients who achieve a response (CR/CRi or PR) may receive itacitinib for up to 8 additional cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of T-cell prolymphocytic leukemia (T-PLL) will be eligible (both treatment naïve and relapsed patients are eligible).
* Age >/= 18 years.
* Patients must not have had chemotherapy or antibody therapy for 7 days prior to starting ITACITINIB. However, patients with rapidly proliferative disease may receive hydroxyurea or decadron until 24 hours prior to starting therapy on this protocol.
* Adequate organ function as defined below: liver function (bilirubin </=2mg/dL, AST and ALT </=3 x ULN or </=5 x ULN if related to leukemic involvement); kidney function (estimated creatinine clearance > 50); known cardiac ejection fraction of > or = 45% within the past 3 months; and platelet count </=30,000.
* ECOG performance status of </= 2.
* A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.

Exclusion Criteria:

* Patients with a diagnosis of T-cell prolymphocytic leukemia (T-PLL) will be eligible (both treatment naïve and relapsed patients are eligible).
* Age >/= 18 years.
* Patients must not have had chemotherapy or antibody therapy for 7 days prior to starting ITACITINIB. However, patients with rapidly proliferative disease may receive hydroxyurea or decadron until 24 hours prior to starting therapy on this protocol.
* Adequate organ function as defined below: liver function (bilirubin </=2mg/dL, AST and ALT </=3 x ULN or </=5 x ULN if related to leukemic involvement); kidney function (estimated creatinine clearance > 50); known cardiac ejection fraction of > or = 45% within the past 3 months; and platelet count </=30,000.
* ECOG performance status of </= 2.
* A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
  The severity of the toxicities will be graded according to the latest version of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). The number and percent of subjects with treatment-emergent adverse events will be summarized according to intensity and drug relationship, and categorized by System Organ Class and preferred term by dose level/Part. All reported AEs that occur after signing informed consent will be included in the analysis of all reported AEs. Exposure to study drug and reasons for discontinuation of study drug will be tabulated. Data will be summarized using descriptive statistics. Continuous variables will be summarized using the number of observations, mean, standard deviation, coefficient of variation, median, and range as appropriate. Categorical values will be summarized using the number of observations and percentages as appropriate.

SECONDARY OUTCOMES:
Response rate (complete remission[CR], complete remission without blood count recovery [CRi], or partial remission [PR]) | Up to 2 years
  The response rate (CR/CRi or PR) will be estimated for all patients along with the 95% confidence interval. Patients with missing or no response assessments will be classified as non-responders. The association between response and patient and clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test. The response rate will be compared between different subgroups (e.g. mutation types) by Fisher exact test.
Duration of response (DOR) | From the first documented onset of PR or CR/CRi to the date of progressive disease/relapse or death due to underlying disease, assessed up to 2 years
  Listed and summarized by the Kaplan-Meier estimator.
Time to response | Up to 2 years
  Listed and summarized by the Kaplan-Meier estimator. Time to response is defined as the time from treatment start till response (CR/CRi/PR) or last follow-up.
Overall survival | From treatment till death or last follow-up, assessed up to 2 years
  Listed and summarized by the Kaplan-Meier estimator.
Event-free survival | From start of treatment to the date of event defined as the first documented progressive disease/relapse, or death due to any cause, whichever comes first, assessed up to 2 years
  Listed and summarized by the Kaplan-Meier estimator. Logrank test will be used to compare the time-to-event difference between different subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kadia TM, Jain A, Rausch CR, Bataller A, Ravandi F, Jabbour E, Qiao W, Borthakur G, Short N, Montalban-Bravo G, Quesada AE, Burger J, Ferrajoli A, Wierda W, Hosing C, Kantarjian H. Phase 1B pilot study of itacitinib with alemtuzumab in patients with T-cell prolymphocytic leukemia. Blood Neoplasia. 2025 Oct 24;3(1):100175. doi: 10.1016/j.bneo.2025.100175. eCollection 2026 Feb. PMID 41536780
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org